CLINICAL TRIAL: NCT06265181
Title: Effect Of Diabetes Coaching on Diabetes Self-Management, Glycoslated Hemoglobin and Diabetes Distress Level in Indıviduals With Type 2 Diabetes: A Randomized Controlled Study
Brief Title: The Effect of Diabetes Coaching on Distress and Diabetes Self-Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Associate Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AIBU-SBF-SK-04
Record Dates: First submitted 2024-02-04; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Coaching; Self Management; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Experimental and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: When the researcher evaluates the participant according to the inclusion criteria, written consent will be obtained from the participant and pre-evaluation forms will be applied when compliance with the criteria is achieved. Afterwards, the participant's group will be notified to the researcher by the independent researcher and randomization will be carried out. With this; Data entries will be made by an independent researcher as group A and group B, without writing the group names. Until the data analysis and reporting is completed, the statistician will be blinded to which group is the intervention and which group is the control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Diabetes coaching will be provided to experimental group participants. In this study, one chemistry interview and eight diabetes coaching meetings are planned to be held.
  Interviews will be conducted in accordance with the standards of the GROW technique, which is based on a scientific framework. Interviews will be held every 10 days, via a video-free phone call, and will last between 45-60 minutes.
  Interventions: Behavioral: Diabetes coaching
- Control Group (No Intervention): Diabetes treatment and care of the participants in this group will continue routinely, and no additional intervention will be performed.

INTERVENTIONS:
Behavioral: Diabetes coaching — Diabetes coaching intervention will be provided to the participants in the intervention group by the researcher, who is a specialist nurse who has received 140 hours of Level 2 Professional Coaching Training and 20 hours of diabetes coaching training. Since each individual's needs and values will be different, diabetes coaching interventions will be tailored specifically to the individual by the researcher within the general coaching framework, but by taking into account the individual's views, awareness, needs and current situation regarding self-management regarding diabetes. This flexibility, which supports the individual-specific approach within the coaching paradigm, is among the key elements in the success of coaching interventions (43). The individual will determine the coaching agenda according to his/her own needs.
  Arms: Intervention Group

SUMMARY:
This research is a randomized controlled, experimental study planned to evaluate the effect of diabetes coaching on diabetes self-management, glycosylated hemoglobin and diabetes distress levels in individuals with type 2 diabetes.

The research is planned to start on 01.01.2024. Participants will be divided into experimental and control groups using the block randomization method. Participants in the experimental group will first receive 8 sessions of diabetes coaching every 10 days after the chemistry interview. No intervention will be made to the control group. The preliminary implementation of the research will be carried out with 4 individuals with diabetes who voluntarily accept participation and meet the inclusion criteria. Data will be collected by face-to-face interview method. Data will be analyzed with IBM SPSS V23 program.

DETAILED DESCRIPTION:
Diabetes is a chronic and metabolic disease that develops when the body cannot secrete enough insulin or the cells cannot use insulin as they should, causing damage to many tissues and organs. It is estimated that there are 537 million adults aged 20-79 in the world with diabetes and this number will reach 783 million in 2045.

Diabetes distress, which is one of the most common mental concerns in individuals with diabetes, makes it difficult to achieve glycemic control, paves the way for the development of diabetes complications and reduces the quality of life. Diabetes distress also causes an increase in the risk of mortality and morbidity. One of the best ways to prevent or reduce diabetes distress is to provide self-management skills and support.

In recent years, health coaching has attracted attention in many countries for improving patients' self-management and providing the necessary behavioral change.

In this study, the effect of coaching intervention applied to individuals with diabetes on diabetes self-management, HbA1c and diabetes distress will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Having been diagnosed with Type 2 diabetes for at least 1 year,
* Being between the ages of 18-65,
* No communication problems,
* Being literate,
* Being able to use a phone (home or mobile phone),
* Lack of diagnosis of psychiatric disease,
* Not receiving hospital treatment due to acute problems,
* Not to be involved in another study involving a similar intervention during the research period

Exclusion Criteria:

* Being diagnosed with type 1 diabetes,
* Type 2 diabetes diagnosis period is less than one year,
* Being under 18 years of age, over 65 years of age,
* Being pregnant,
* Having a diagnosis of psychiatric disease,
* Not agreeing to participate in the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-03-27 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Type 2 Diabetes Self-Management Scale | 3 months
  This scale was developed by Koç and Özkan to evaluate self-management in type 2 diabetics and is a 5-point Likert type ("Always=5", "Often=4", "Sometimes=3") , "Rarely=2", "Never=1"). The sub-dimensions of the scale, which consists of a total of 19 questions; "Healthy Lifestyle Behaviors" (11 items), "Use of Health Services" (4 items) and "Blood Sugar Management" (4 items). The highest score that can be obtained from the scale is 95 and the lowest score is 19. As the score obtained from the scale increases, diabetes self-management increases. The Cronbach alpha value of the scale was calculated as 0.856 (37)

SECONDARY OUTCOMES:
Diabetes Distress Scale | 3 months
  The Diabetes Distress Scale is a 17-item, 6-point Likert type scale developed by Polonsky et al. in 2005 to evaluate diabetes-specific distress. The scale consists of four subscales: emotional burden, doctor-related distress, treatment-related distress, and interpersonal distress. Each question in the scale is scored between 1 point and 6 points, and the scale evaluates the distress experienced by the individual in the last month (40). The validity and reliability study of the scale was conducted by Çakıllı et al. in 2015, and the α value was found to be 0.88 for the entire scale and 0.90 for each of the subscales. The average total score of the scale is calculated by dividing the total score of the answers given to the scale by 17. A score of 3 points or higher suggests the presence of distress. Score calculation for the sub-dimensions is obtained by dividing the total score of the answers given to the questions by the number of questions in that section (40,41)
HbA1c Monitoring Form | 3 months
  This is the form created to monitor the HbA1c values of individuals with diabetes before and after the application and to follow the changes (Annex 3). HbA1c is a routine test evaluated every three months in the follow-up of individuals with diabetes. Individuals will be included in the study if they have HbA1c tests within the last 10 days when they come to the Family Health Care, otherwise they will be included in the study when they have the test done on a date suitable for routine control.
Introductory Features Form | 3 months
  The form was prepared by the researcher by conducting a literature review and consists of a total of 23 questions (32,34,37-39). In this form, in the first section; Questions about age, gender, education level, marital status, perceived income level, who the individual lives with, smoking and alcohol use, and the presence of chronic diseases. In the second part, there are questions about diabetes; duration of diabetes diagnosis, type of diabetes treatment, status of receiving diabetes education, HbA1c value measured in the last 10 days, presence and types of complications due to diabetes, regular use of diabetes medications, how diabetes care is carried out, status of receiving diabetes education (from whom, training subject , when it was taken, etc.) are included

CONTACTS AND LOCATIONS:
Overall Officials: Saadet CAN ÇİÇEK, Assoc Prof., Principal Investigator — Abant Izzet Baysal University

IPD SHARING:
Plan to Share IPD: No